CLINICAL TRIAL: NCT01443676
Title: Avastin Plus Radiotherapy in Elderly Patients With Glioblastoma
Acronym: ARTE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARTE
Record Dates: First submitted 2011-08-12; First posted 2011-09-30 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Glioblastoma
MeSH Terms: conditions — Glioblastoma | interventions — Bevacizumab; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Radiotherapy (Active Comparator): Radiotherapy
  Interventions: Radiation: Radiation therapy
- Radiotherapy plus Bevacizumab (Experimental): Radiotherapy plus Bevacizumab
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Bevacizumab will be added to radiotherapy
  Other Names: Avastin
  Arms: Radiotherapy plus Bevacizumab
Radiation: Radiation therapy — Radiation therapy
  Arms: Radiotherapy

SUMMARY:
The purpose of this study is to explore the efficacy of bevacizumab combined with radiotherapy compared with radiotherapy alone in the treatment of newly diagnosed glioblastoma in the elderly.

* Trial with medicinal product

DETAILED DESCRIPTION:
This is a randomized (2:1), explorative, parallel-group, open-label, phase II trial in elderly patients with newly diagnosed glioblastoma. In the control arm, patients will receive radiotherapy, in the experimental arm, patients will receive bevacizumab during and after radiotherapy until progression.

Background:

For decades, neurosurgical resection and postoperative radiotherapy have been the cornerstones of treatment for patients with glioblastoma. Most chemotherapeutic agents showed little or no activity in malignant glioma patients, with the possible exception of nitrosoureas. This has changed with the introduction of temozolomide, first shown to be active in recurrent disease (Yung et al. 2000) and more recently in newly diagnosed glioblastoma (Stupp et al. 2005, 2009). This EORTC 26981-22981 NCIC CE.3 trial demonstrated an increase in median survival from 12.1 to 14.6 months and of the 2 year survival rate from 10% to 26% in patients receiving radiotherapy plus temozolomide compared with radiotherapy alone. Notably patients with tumors exhibiting methylation of the promoter region of the O6-methylguanine DNA methyltransferase (MGMT) gene showed a striking benefit from temozolomide (Hegi et al. 2005). Yet, inclusion in this trial was limited to patients up to the age of 70, and subgroup analyses demonstrated that younger patients were more likely to derive benefit from combined modality treatment than older patients. Thus, radiotherapy alone is still the standard of care in the elderly. The value of radiotherapy has been confirmed in a small randomized trial comparing best supportive care versus radiotherapy alone: median survival was 29 weeks with radiotherapy compared with 16.9 weeks with supportive care only (Keime-Guibert et al. 2007). Based on the overall shorter survival in elderly patients, hypofractionated radiotherapy has been explored and shown to be equieffective in patients aged 65-70 years and more (Roa et al. 2004). Two randomized trials presented in abstract form at the Annual Meeting of the American Society of Clinical Oncology in June 2010 failed to show superiority of primary temozolomide chemotherapy alone over radiotherapy alone in elderly patients (Malmstrom et al. 2010, Wick et al. 2010a). In fact, the German NOA-08 trial even showed that primary temozolomide alone is not non-inferior to primary radiotherapy alone (Wick et al. 2010a). A concomitant treatment strategy is currently evaluated in a NCIC-EORTC randomized trial. Further, the Nordic trial corroborated the equieffectiveness of an accelerated radiotherapy protocol of 40 Gy administered in 15 fractions versus the standard fractionation of 30 x 2 Gy. Altogether, these clinical data justify the exploration of new, temozolomide-free first-line treatment strategies in glioblastoma.

Glioblastomas express high levels of vascular endothelial growth factor (VEGF) and are highly vascularized tumors. The VEGF antibody, bevacizumab, has recently gained approval in patients with recurrent glioblastoma in the USA and in Switzerland in 2009, but not in the EU. Its role in the first-line treatment of glioblastoma is currently being evaluated in randomized trials. There is limited data on the safety and efficacy of bevacizumab in elderly patients with glioblastoma, although the safety profile of bevacizumab in elderly patients with other types of cancer, e.g., lung cancer is favorable. There are ample rationales for combining bevacizumab with radiotherapy, including the induction of VEGF by radiotherapy and the concept of vascular normalization resulting in increased oxygenation and thus sensitivity to radiotherapy. Thus, bevacizumab is not only expected to inhibit angiogenesis, but may also exhibit additive or synergistic interactions with radiotherapy and further impair tumor growth. Altogether, this study seeks to explore, using a dedicated neuroimaging protocol, the possibility that bevacizumab enhances the effects of radiotherapy via the process of vascular normalization.

The purpose of this study is to explore the efficacy of bevacizumab combined with radiotherapy compared with radiotherapy alone in the treatment of newly diagnosed glioblastoma in the elderly.

ELIGIBILITY:
Inclusion criteria: Diagnosis: newly diagnosed glioblastoma in elderly patients

1. Signed informed consent
2. Age > 65 years
3. Newly diagnosed supratentorial glioblastoma
4. Eligible for first infusion of bevacizumab > 28 and > 49 days after surgery for glioblastoma
5. Karnofsky performance score 60 or more
6. Paraffin-embedded tissue for central pathology review
7. Stable or decreasing corticosteroid dose within 5 days prior to enrolment
8. Adequate haematological function:
9. Adequate liver function
10. Adequate renal function

Exclusion criteria:

1. Karnofsky performance score 50 or less
2. Evidence of recent hemorrhage on postoperative brain MRI
3. Tumor with infiltration of retina, optic nerve, optic chiasm or brainstem
4. Any prior chemotherapy including carmustine-containing wafers (Gliadel®) or immunotherapy for glioblastoma or lower grade astrocytomas
5. Any prior radiotherapy to the brain or prior radiotherapy resulting in a potential overlap in the radiation field
6. Inadequately controlled hypertension
7. History of hypertensive crisis or hypertensive encephalopathy
8. New York Heart Association (NYHA) grade II or higher congestive heart failure
9. Myocardial infarction or unstable angina within 6 months prior to enrolment
10. Stroke or transitory ischemic attack within 6 months prior to enrolment
11. Other significant vascular disease within 6 months prior to enrolment
12. History of = grade 2 haemoptysis within 1 month prior to enrolment
13. Bleeding diathesis or coagulopathy in the absence of therapeutic anticoagulation
14. Major surgical procedure, open biopsy, intracranial biopsy, ventriculoperitoneal shunt or significant traumatic injury within 28 days prior to first dose of bevacizumab
15. Core biopsy (excluding intracranial biopsy) or other minor surgical procedure within 7 days prior to first dose of bevacizumab
16. Abdominal fistula or gastrointestinal perforation within 6 months prior to enrolment
17. Intracranial abscess within 6 months prior to enrolment
18. Serious non-healing wound, active ulcer or untreated bone fracture
19. Pregnancy or lactation
20. Fertile women < 2 years after last menstruation and men unwilling or unable to use effective means of contraception
21. Active malignancy that may interfere with the study treatment at the investigator?s and PI discretion

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 75 (Actual)
Dates: Start 2011-10; Primary Completion 2015-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
median overall survival | 1 year
  median overall survival

SECONDARY OUTCOMES:
progression-free survival | progression-free survival after 6 months
  progression-free survival after 6 months

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich; Michael Weller, Professor, Principal Investigator — University Hospital Zurich, Division of Neurology
Locations (1):
- Department of Neurology, University Hospital Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Wirsching HG, Roelcke U, Weller J, Hundsberger T, Hottinger AF, von Moos R, Caparrotti F, Conen K, Remonda L, Roth P, Ochsenbein A, Tabatabai G, Weller M. MRI and 18FET-PET Predict Survival Benefit from Bevacizumab Plus Radiotherapy in Patients with Isocitrate Dehydrogenase Wild-type Glioblastoma: Results from the Randomized ARTE Trial. Clin Cancer Res. 2021 Jan 1;27(1):179-188. doi: 10.1158/1078-0432.CCR-20-2096. Epub 2020 Sep 23. PMID 32967939
- [Derived] Wirsching HG, Tabatabai G, Roelcke U, Hottinger AF, Jorger F, Schmid A, Plasswilm L, Schrimpf D, Mancao C, Capper D, Conen K, Hundsberger T, Caparrotti F, von Moos R, Riklin C, Felsberg J, Roth P, Jones DTW, Pfister S, Rushing EJ, Abrey L, Reifenberger G, Held L, von Deimling A, Ochsenbein A, Weller M. Bevacizumab plus hypofractionated radiotherapy versus radiotherapy alone in elderly patients with glioblastoma: the randomized, open-label, phase II ARTE trial. Ann Oncol. 2018 Jun 1;29(6):1423-1430. doi: 10.1093/annonc/mdy120. PMID 29648580